CLINICAL TRIAL: NCT01095952
Title: Reduction of Ventricular Rate During Atrial Fibrillation by AV Node Stimulation" AVNS Download Study
Brief Title: AV-node Stimulation Clinical Download Study to Reduce Ventricular Rate During AF
Acronym: AVNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic BRC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVNS
Record Dates: First submitted 2010-03-11; First posted 2010-03-30 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; inappropriate shock; AV-node stimulation; ventricular arrhythmia
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AVNS ON (Experimental): Consulta downloaded with AVNS to provide high frequency bursting during fastly conducted AF. AVNS will be programmed on for five months. The feasibility and safety of the AVNS algorithm to reduce inappropriate shocks will be monitored.
  Interventions: Device: AVNS ON

INTERVENTIONS:
Device: AVNS ON — Delaying the AV-node by stimulating the parasympathetic nerves innervating the AV-node with high frequency burst pacing during the refractory period of the ventricle using a standard atrial lead at a septal position.
  Other Names: AVNS; AV-node stimulation; parasympathetic AV-node stimulation

SUMMARY:
The aim of this multi-center research study is to evaluate the performance (primary purpose) and safety of a new algorithm aimed at controlling ventricular rate (VR) during rapidly conducted atrial fibrillation (AF) by delivering AV node stimulation (AVNS) from the atrial lead placed at a septal position, and designed with the purpose of reducing inappropriate shocks. Additional purposes include the assessment of a possible application of AVNS aimed at allowing prolonged control of VR during AF and reducing AF symptoms, and evaluation of implantation data on selective placement of the atrial lead in postero-septal right atrium. About 37 patients will be followed for half a year.

DETAILED DESCRIPTION:
The aim of this multi-center research study is to evaluate the performance (primary purpose) and safety of a new algorithm aimed at controlling VR during rapidly conducted AF by delivering AVNS from the atrial lead placed at a septal position, and designed with the purpose of reducing inappropriate shocks. Additional purposes include the assessment of a possible application of AVNS aimed at allowing prolonged control of VR during AF and reducing AF symptoms, and evaluation of implantation data on selective placement of the atrial lead in postero-septal right atrium. About 37 patients will be followed for half a year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a documented history of paroxysmal or persistent AF are eligible to be enrolled in the study if one of the following criteria is met:
* Indication for CRT implant according to current Guidelines (Heart Failure, NYHA III-IV class, symptomatic despite optimal stable medical therapy, left ventricular (LV) ejection fraction ≤35% and QRS≥120ms); OR
* Indication for upgrading to CRT-D from a single chamber device; OR
* Indication for upgrading to CRT-D from a dual chamber device with septal atrial lead or a dislodged atrial lead; OR
* Indication for device replacement or surgical revision in patients already implanted with a CRT-D device and an atrial lead in the septal position or a dislodged atrial lead; OR
* Patients already implanted with a ConsultaTM device and an atrial lead in the septal position, requiring electrical cardioversion.

Exclusion Criteria:

* If any of the following criteria are met, patient cannot be enrolled in the study:
* Permanent atrial fibrillation;
* Patients who are not on anti-coagulant therapy;
* Advanced AV block (II-III degree AV block);
* Patients previously submitted to valvular surgery;
* Patients previously submitted to AV or AF ablative procedures;
* Age < 18 years;
* Patient not disposed to sign the Informed Consent;
* Participation in other studies which could potentially conflict with this study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the performance of the investigational algorithm in reducing mean VR during AF, the relative reduction of VR during AVNS will be assessed in acute in-hospital tests, conducted preferably during either spontaneous or induced episodes of AF. | baseline and 1 month

SECONDARY OUTCOMES:
To evaluate the performance of the investigational algorithm in shock reduction. | baseline, 1 month, 3 months, 6 months
  assessing the number of successful rate reduction interventions by AVNS during spontaneous episodes of AF occurring during follow-up, with rapid VR due to AF conducted in the VT/FVT/VF zone;
To evaluate the safety of the investigational algorithm. | baseline, 1 month, 3 months, 6 months
  To evaluate the safety of the investigational algorithm, assessing:
  * The rate of adverse device effects and serious adverse device effects related to the investigational algorithm;
  * The number of VT/VF or AT/AF episodes potentially induced or prolonged by the investigational algorithm.
To gather data for further possible applications. | baseline, 1 month, 3 months, 6 months
  To gather data for further possible applications of AVNS, assessing:
  * the performance of the investigational algorithm in decreasing mean VR and standard deviation directly after 30 seconds of AVNS as compared to 30 seconds directly before algorithm intervention (baseline: all patients; 1, 3 and 6 months follow-up: patients in AF only);
  * the performance of the investigational algorithm in combination with ventricular pacing in decreasing mean VR and standard deviation directly after 30 seconds of AVNS as compared to 30 seconds directly before algorithm intervention (baseline only).
To collect data on selective placement of the atrial lead. | baseline, 1 month, 3 months, 6 months
  evaluating:
  * electrical characteristics (impedance, threshold, sensing, FFRW) related to pacing and AVNS at implant (when applicable), baseline and follow-ups;
  * the percentage of atrial lead implantations with electrical characteristics suitable both for standard pacing and AVNS;
  * adverse events related to selective atrial lead placement at implant and in the follow-up;
  * mean duration of implant procedure and mean fluoroscopic time;
  * the presence of an implant learning curve.

CONTACTS AND LOCATIONS:
Overall Officials: Stephano Bianchi, MD, Principal Investigator — Department of Cardiology, Hospital Rome, ospedalis giovanni calibita fatebenefratelli
Locations (4):
- Klinikum Aachen, Aachen, Germany
- Italy (2):
  - Institute of Internal Medicine and Cardiology, Firenze, Florence
  - Department of Cardiology, Ospedalis Giovanni Calibita Fatebenefratelli, Rome, Rome
- Department of Cardiology, University Hospital, Uppsala, Sweden

REFERENCES:
- [Background] Bianchi S, Rossi P, Della Scala A, Kornet L, Pulvirenti R, Monari G, Di Renzi P, Schauerte P, Azzolini P. Atrioventricular (AV) node vagal stimulation by transvenous permanent lead implantation to modulate AV node function: safety and feasibility in humans. Heart Rhythm. 2009 Sep;6(9):1282-6. doi: 10.1016/j.hrthm.2009.05.011. Epub 2009 May 9. PMID 19716083
- [Background] Rossi P, Bianchi S, Barretta A, Della Scala A, Kornet L, De Paulis R, Bellisario A, D'Addio V, Pavaci H, Miraldi F. Post-operative atrial fibrillation management by selective epicardial vagal fat pad stimulation. J Interv Card Electrophysiol. 2009 Jan;24(1):37-45. doi: 10.1007/s10840-008-9286-2. Epub 2008 Aug 30. PMID 18758932
- [Background] Bianchi S, Rossi P, Della Scala A, Kornet L. Endocardial transcatheter stimulation of the AV nodal fat pad: stabilization of rapid ventricular rate response during atrial fibrillation in left ventricular failure. J Cardiovasc Electrophysiol. 2009 Jan;20(1):103-5. doi: 10.1111/j.1540-8167.2008.01243.x. Epub 2008 Jul 3. PMID 18631264
- [Derived] Bianchi S, Rossi P, Schauerte P, Elvan A, Blomstrom-Lundqvist C, Kornet L, Gal P, Mortsell D, Wouters G, Gemein C. Increase of ventricular interval during atrial fibrillation by atrioventricular node vagal stimulation: chronic clinical atrioventricular-nodal stimulation download study. Circ Arrhythm Electrophysiol. 2015 Jun;8(3):562-8. doi: 10.1161/CIRCEP.114.002588. Epub 2015 Apr 15. PMID 25878323